CLINICAL TRIAL: NCT05679856
Title: Vocal Cord Only Hypofractionated Radiotherapy vs Whole Laryngeal Radiotherapy for T1aN0 Glottic Cancer
Brief Title: Vocal Cord vs Whole Laryngeal Radiotherapy for T1aN0 Glottic Cancer
Acronym: VC-Larynx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R02002-30908
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Larynx Cancer Stage I; Glottic Carcinoma
Keywords: Larynx; Glottic; T1; hypofractionated radiotherapy; Vocal cord; Laryngeal carcinoma
MeSH Terms: conditions — Laryngeal Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Single vocal cord hypofractionated radiotherapy (Experimental): Hypofractionated radiotherapy 58.08Gy/16 fractions to affected vocal cord plus margins to account for motion and setup errors using IMRT/VMAT technique
  Interventions: Radiation: Hypofractionated single vocal cord irradiation
- Whole laryngeal radiotherapy (Active Comparator): Radiotherapy 63Gy/28 fractions to whole larynx from lower border of hyoid bone to lower border of cricoid cartilage using IMRT/VMAT technique
  Interventions: Radiation: Whole laryngeal radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated single vocal cord irradiation — Only the affected vocal cord with additional margin to account for motion and setup errors will receive 58.08Gy/16 fractions using IMRT/VMAT technique
  Arms: Single vocal cord hypofractionated radiotherapy
Radiation: Whole laryngeal radiotherapy — The whole larynx from lower border of hyoid bone to lower border of cricoid cartilage will receive 63Gy/28 fractions using IMRT/VMAT technique
  Arms: Whole laryngeal radiotherapy

SUMMARY:
The primary objective of this prospective randomized clinical trial is to assess non inferiority in terms of local control achieved with single vocal cord hypofractionated radiotherapy compared to standard of care whole laryngeal radiotherapy in patients with T1aN0 glottic cancer . Secondary objectives include overall survival rate and to compare the Voice Handicap Index score between the 2 arms as well as acute and late toxicities. Patients are randomized in 1:1 ratio.

DETAILED DESCRIPTION:
Most laryngeal cancers present in early stage and more than two thirds of it occur in the glottic region(T1-T2). Early glottic carcinoma is historically treated with conventional radiotherapy using large box fields (from lower border of hyoid to lower border of cricoid), using wedged parallel opposed photon beams. In spite of good local control rate of more than 90% for T1a glottic cases, the tumor-free contralateral vocal cord, arytenoids, thyroid cartilage, and all muscles responsible for opening and closing the vocal cords, the swallowing muscles, carotid arteries and thyroid gland are exposed to high radiation doses (fully or partially) which could lead to an increased probability of complications that negatively influence the quality of life of these patients. Typical complications have involved voice/ speech impairment, diet problems (swallowing, trismus), arytenoids edema, an increased risk of strokes, and reduced treatment options for previously irradiated patients. Many studies showed that increasing fraction size and shortening the overall treatment time (hypofractionated radiotherapy) could result in better local control of T1 glottic cancer The use of 63Gy/28 Fractions(Fx) showed superior local control compared with conventional use of 66Gy/33Fx with shorter overall treatment time. Based on this study this dose is the standard in our institute. In contrast to the traditional radiotherapy principle to treat the whole larynx, surgical laser excision of T1a glottic cancer involves removal of gross tumor with minimal, often sub-millimeter, excisional margins with good oncological outcome and good quality of voice. Similar to this surgical concept and with modern radiotherapy IMRT/VMAT technique, the approach of single vocal cord irradiation (SVCI) was introduced. A study of 30 patients with T1a glottis cancer treated by image guided vocal cord radiotherapy was published in 2015 and it showed 100% local control at 2 years and with no grade 3 toxicities reported and better quality of voice when compared to historical cohorts Dosimetric analysis showed that IMRT resulted in markedly reducing the dose to contralateral cord, arytenoids, thyroid cartilage, inferior constrictor muscle and carotid arteries. To date no prospective phase 3 trial was done to compare treatment outcome and toxicity profile of vocal cord only hypofractionated radiotherapy vs traditional whole laryngeal radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* T10N0 glottic squamous cell carcinoma
* Ability to provide written informed consent
* Eastern Cooperative Oncology Group performance status 0-2

Exclusion Criteria:

* Previous head and neck irradiation.
* WHO performance status above 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Local control | at 1 year follow up
  Rate of local control

SECONDARY OUTCOMES:
Voice Handicap index | Pretreatment- 2 months 6 months 1 year and 1 year follow upn
  Voice Handicap index score Scores are rated on a 0-4 scale to indicate the presence and severity of the symptoms. Lower scores represent better functioning and quality of life.
Rates of acute toxicity | Week 0 post-treatment and at 2-month follow-up
  Rates of acute toxicity as per CTCAE v5.0
Rates of chronic toxicity | at 6 months - 1 year and 2 years follow up
  Rates of chronic toxicity as per CTCAE v5.0
Overall survival | at 2 year follow up
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mortada Elsharief, Principal Investigator — NCI, Cairo University, Egypt; Tarek Shouman, Study Chair — NCI, Cairo University, Egypt
Locations (1):
- National Cancer Institute, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamazaki H, Nishiyama K, Tanaka E, Koizumi M, Chatani M. Radiotherapy for early glottic carcinoma (T1N0M0): results of prospective randomized study of radiation fraction size and overall treatment time. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):77-82. doi: 10.1016/j.ijrobp.2005.06.014. Epub 2005 Sep 19. PMID 16169681
- [Background] Gowda RV, Henk JM, Mais KL, Sykes AJ, Swindell R, Slevin NJ. Three weeks radiotherapy for T1 glottic cancer: the Christie and Royal Marsden Hospital Experience. Radiother Oncol. 2003 Aug;68(2):105-11. doi: 10.1016/s0167-8140(03)00059-8. PMID 12972304
- [Background] Al-Mamgani A, Kwa SL, Tans L, Moring M, Fransen D, Mehilal R, Verduijn GM, Baatenburg de Jong RJ, Heijmen BJ, Levendag PC. Single Vocal Cord Irradiation: Image Guided Intensity Modulated Hypofractionated Radiation Therapy for T1a Glottic Cancer: Early Clinical Results. Int J Radiat Oncol Biol Phys. 2015 Oct 1;93(2):337-43. doi: 10.1016/j.ijrobp.2015.06.016. Epub 2015 Jun 14. PMID 26264629
- [Background] Osman SO, Astreinidou E, de Boer HC, Keskin-Cambay F, Breedveld S, Voet P, Al-Mamgani A, Heijmen BJ, Levendag PC. IMRT for image-guided single vocal cord irradiation. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):989-97. doi: 10.1016/j.ijrobp.2010.12.022. Epub 2011 Feb 6. PMID 21300449
- [Background] Dornfeld K, Simmons JR, Karnell L, Karnell M, Funk G, Yao M, Wacha J, Zimmerman B, Buatti JM. Radiation doses to structures within and adjacent to the larynx are correlated with long-term diet- and speech-related quality of life. Int J Radiat Oncol Biol Phys. 2007 Jul 1;68(3):750-7. doi: 10.1016/j.ijrobp.2007.01.047. Epub 2007 Apr 6. PMID 17418971